CLINICAL TRIAL: NCT04958681
Title: Changes in Physical Activity Status: Comparison of Older Adults With Versus Without a History of Covid-19 Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Bilal Katipoglu, Divsion of Geriatric, Gulhane Training and Research Hospital
Other Study IDs: 2020-305
Record Dates: First submitted 2021-07-07; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Covid19
Keywords: physical activity
MeSH Terms: conditions — COVID-19; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 history positive
  Interventions: Other: exercise
- Covid-19 history negative
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — The participants were subsequently asked whether the pandemic had altered their physical activity status and rate the severity of reduction in mobility level compared to the period before the Covid-19 with the following options: none, 0; mild, 1; moderate, 2; severe, 3. Then, the participants were also asked whether they perform a physical exercise in a home setting. We recorded regular outdoor physical activity and home-based exercises (only after the pandemic) as a dichotomous variable (yes or no). The number of physical activity days per week was also obtained.

SUMMARY:
The negative impact of the Covid-19 pandemic on the physical activity behavior of overall adults has been reported. But much less is known in older adults. Alterations in physical activity among Covid-19 survivors have not been investigated so far. The present study aimed to evaluate the physical activity status of older adults in terms of a history of Covid-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* 65 years non-dementia community dwelling older adults

Exclusion Criteria:

* The exclusion criteria were: (1) intensive care unit admission due to Covid-19 infection, (2) neurodegenerative or psychotic disease, (3) delirium, (4) terminal illness (malignancy, advanced organ failure), and (5) hearing impairment that disrupts conducting the telephone survey

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The patients were matched with a control group of 76 community-dwelling older individuals without a Covid-19 diagnosis in the same period.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-07-21 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-09-11 (Estimated)

PRIMARY OUTCOMES:
physical activity | 1 year fellow-up
  telephone based questionare related to frequency and duration of phyiscal activity

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane training and research hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No